CLINICAL TRIAL: NCT05096000
Title: InterMob: a Randomized Controlled Trial Aimed at Reducing Car Use in Regular Car Users by Combining Hard and Soft Levers
Brief Title: InterMob: a Randomized Controlled Trial Aimed at Reducing Car Use in Regular Car Users
Acronym: InterMob
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Aina Chalabaev (Other)
Collaborators: IDEX - Univ. Grenoble-Alpes (Unknown); Région Auvergne-Rhône Alpes (Unknown); Institut de Recherche en Santé Publique, France (Other); ADEME (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Métropole Grenoble-Alpes (Unknown)
Responsible Party: Sponsor-Investigator, Aina Chalabaev, Professor, Université Joseph Fourier
Organization: Université Joseph Fourier (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INTERMOBFRUGA
Record Dates: First submitted 2021-09-22; First posted 2021-10-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Automobile Driving; Active Commuting
Keywords: Transportation; Active transportation; Sustainable transportation; physical activity; air pollution
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the participants nor the outcomes assessors will know the intervention in which each participant is assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- InterMob: a behavioral and economical intervention (Experimental): * 6 months of free transport/bicycle (12.5 Adding objects in the BCT, Michie et al., 2011)
  * Two meetings with a coach :
    1. st meeting: discussion about the motivations to change (motivational interviewing and 5.2 Salience of consequences, BCT), personalized advice of transport (4.1 Instruction on how to perform the behavior, BCT), mobility change goals, and action planning (1.1 Goal setting and 1.4 Action planning, BCT), solutions to possible obstacles (1.2 Problem solving, BCT)
    2. nd meeting: discussion about the goals and the obstacles lived and resolved. If needed, personalized transport advice is given.
  * "Goals notebook" to fill up for 6 months (goals need to be set every 2 weeks and obstacles if experienced)
  * Weekly SMS during 6 months, prompting a) to set and adapt goals (1.7 Review outcome, BCT) and b) to do a self-feedback related to mobility change (e.g. a more important well-being) (2.4 Self-monitoring of outcomes, BCT's taxonomy)
  Interventions: Behavioral: InterMob: a randomized controlled trial aimed at reducing car use in regular car users
- Air pollution information: an informational group (Other): Active control group focused on air pollution information:
  * Two meetings with a coach:
    1. st meeting: Discussion about air pollution (definition, sources, population most affected, levels in Grenoble, the consequences on health, pollution peaks), air pollution and car use (video about the pollution exposure of car drivers and the consequences of fine particles) and, a discussion about the benefit and disadvantages of using a car (5.2 Salience of consequences according to BCT's taxonomy)
    2. nd meeting: Discussion about air quality during the last weeks and they check the quality of air of the last week.
  * "Observation notebook" to fill up for 6 months (quality of air in Grenoble and the pollution peaks every 2 weeks)
  * Weekly SMS during 6 months prompting a) to write down the air quality of the air every two weeks and b) write down any pollution peak announced in the television/radio/telephone
  Interventions: Other: Active control: Air pollution information

INTERVENTIONS:
Behavioral: InterMob: a randomized controlled trial aimed at reducing car use in regular car users — Intermob is a theory- and evidence-based behavioral intervention that combines public transport/bicycle and motivational techniques (action planning, personalized transport advice, goal setting).
  Arms: InterMob: a behavioral and economical intervention
Other: Active control: Air pollution information — The active control intervention is based on a discussion about air pollution, the effects of air pollution on health, the association between air pollution and transport.
  Arms: Air pollution information: an informational group

SUMMARY:
Regular car use is a source of pollution and physical inactivity. InterMob is an interdisciplinary randomized controlled behavioral intervention aiming at reducing car use. The objectives of InterMob are to a) Evaluate the efficacy of a theory- and evidence-based intervention, b) Identify the mechanisms related mobility change, and c) Identify the conditions under which the intervention is effective.

To meet these objectives, 300 regular car users living in Grenoble will be recruited and randomized in one of two arms:

1. experimental group that will receive the InterMob intervention: six months of free public transport/access to a bicycle, and behavior change techniques (personalized transport advice, setting of mobility change goals, considering possible obstacles; 6 months of motivational messages to prompt goal setting and self-monitoring).
2. active control group that will receive information about air pollution (discussion about the health consequences of air pollution, the association between air pollution and car use; 6 months of messages to prompt air pollution monitoring.) Follow-up measures will be carried out until 24 months after the beginning of the study (8-day measurement sessions). Five sessions will involve wearing a GPS/accelerometer, and an air pollution sensor. Participants will complete mobility logs and questionnaires measuring the psychological mechanisms related to their mobility (habits, intentions, self-efficacy), and socio-economical characteristics (number of children, accessibility) during the 8 sessions.

The investigators hypothesize that the participants allocated to experimental group will reduce the car use and increase the use of alternative modes to the car (biking, walking, public transport, and carpooling) more than the participants of the control group, and that these changes will remain. The investigators hypothesize that mobility changes will be mediated by intention and self-efficacy. The investigators hypothesize that the efficacy of the intervention will be moderated by socio-spatial factors (number of children, travel distances) and psychological factors (self-control).

The main criterion will be car use reduction and the use of alternative modes to the car. In addition, the investigators will assess physical activity (minutes of moderate-to-vigorous physical activity), the exposure to air pollution, the quality of life and the carbon footprint associated to transport.

DETAILED DESCRIPTION:
Sample size : The investigators have calculated the sample size considering :

* the proportion of trips made by car (49% of the trips made in Grenoble Metropole are made by car according to the EMD, 2010 which is the most recent survey in the area currently available),
* the potential target population's transport behavior (a percentage of the population can be classified as reluctant drivers with positive attitudes toward other modes of transportation, this population makes 80% of their trips and could potentially reduce their car use to 64% considering the characteristics of the trips)
* the impact of past interventions (car reduction of -17%, from 50% to 33% of car use, Brockman & Fox, 2011).

The investigators considered a statistical power of 0.8, and a significance level of 0.05 for a proportion of 80% or 50% of trips made by car in the control group. In order to detect a difference of 15% when the share of trips made by car is reduced from 80% to 65% or from 50 to 35%, the investigators need 300 individuals (i.e., 150 individuals in each group).

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old at the time of inclusion

  • Profile: employed / unemployed / retired / on work-study or apprenticeship
  * If employed : Work and live in the SMAAG territory (Metropole of Grenoble + Grésivaudan + Pays voironnais)
  * If in apprenticeship/training program: Working, studying and living in the SMAAG territory (Metropole of Grenoble + Grésivaudan + Pays voironnais)
  * If unemployed / retired : Reside in the SMAAG territory (Metropole of Grenoble + Grésivaudan + Pays voironnais)
* The car/motorcycle/scooter is the main mode of travel during the week (excluding weekends)
* Travels 3, 4, or 5 days by car (excluding weekdays)
* Thinks about reducing car use or has started to reduce car use - Expect to live and work in the Grenoble area in the next 2 years (Very likely and likely options)

Exclusion Criteria:

* Being a student
* Living outside the Metropole of Grenoble + Grésivaudan + Pays voironnais
* Working outside (Metropole of Grenoble + Grésivaudan + Pays voironnais)
* Studying outside (Metropole of Grenoble + Grésivaudan + Pays voironnais)
* Car/motorcycle/scooter is not the main mode of travel
* Travels 0, 1 or 2 days a week by car
* Does not intend to reduce the frequency of car use
* Does not expect to live and/or work in the Grenoble area in the next 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in car use from the baseline and the beginning of the intervention (one month after the beginning of the intervention, Month 1) | Baseline and one month and a half after the baseline (Month 1)
  Car use (kilometers traveled and modal share) will be measured using the GPS tracks collected by a GPS device (SenseDoc) and by calculating the variables of interest from the information mentioned in the travel diary. The GPS device is used during 9 days each and the travel diary is filled up during 8 days
Changes in car use from the baseline and half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  Car use (kilometers traveled and modal share) will be measured using the GPS tracks collected by a GPS device (SenseDoc) and by calculating the variables of interest from the information mentioned in the travel diary. The GPS device is used during 9 days each and the travel diary is filled up during 8 days
Changes in car use from the baseline the end of the intervention (Month 7) | Baseline and seven months after the baseline (Month 7)
  Car use (kilometers traveled and modal share) will be measured using the GPS tracks collected by a GPS device (SenseDoc) and by calculating the variables of interest from the information mentioned in the travel diary. The GPS device is used during 9 days each and the travel diary is filled up during 8 days
Changes in car use from the baseline and two months after the end of the intervention (Month 9) | Baseline and nine months after the baseline (Month 9)
  Car use (kilometers traveled and modal share) will be measured by calculating the variables of interest from the information mentioned in the travel diary. Travel diary is filled up during 8 days
Changes in car use from the baseline and six months after the end of the intervention (Month 12) | Baseline and one year after the baseline (Month 12)
  Car use (kilometers traveled and modal share) will be measured by calculating the variables of interest from the information mentioned in the travel diary. Travel diary is filled up during 8 days
Changes in car use from the baseline and one year after the end of the intervention (Month 18) | Baseline and one year and a half after the baseline (Month 18)
  Car use (kilometers traveled and modal share) will be measured using the GPS tracks collected by a GPS device (SenseDoc) and by calculating the variables of interest from the information mentioned in the travel diary. The GPS device is used during 9 days each and the travel diary is filled up during 8 days
Changes in car use from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline and two years after the baseline (Month 24)
  Car use (kilometers traveled and modal share) will be measured by calculating the variables of interest from the information mentioned in the travel diary. Travel diary is filled up during 8 days

SECONDARY OUTCOMES:
Changes in active commuting (classic or electric bike, public transport, walk, carpooling) from the baseline and and the beginning of the intervention (one month after the beginning of the intervention, Month 1) | Baseline and one month and a half after the baseline (Month 1)
  Active commuting will be measured using the GPS tracks and by calculating the variables of interest from travel diary (kilometers traveled, modal share). The GPS device is used during 9 days each and the travel diary is filled up during 8 days.
Changes in active commuting (classic or electric bike, public transport, walk, carpooling) from the baseline and the half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  Active commuting will be measured using the GPS tracks and by calculating the variables of interest from travel diary (kilometers traveled, modal share). The GPS device is used during 9 days each and the travel diary is filled up during 8 days.
Changes in active commuting (classic or electric bike, public transport, walk, carpooling) from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Active commuting will be measured using the GPS tracks and by calculating the variables of interest from travel diary (kilometers traveled, modal share). The GPS device is used during 9 days each and the travel diary is filled up during 8 days.
Changes in active commuting (classic or electric bike, public transport, walk, carpooling) from the baseline and two months after the end of the intervention (Month 9) | Baseline, and nine months after the baseline (Month 9)
  Active commuting will be measured by calculating the variables of interest from travel diary (kilometers traveled, modal share). The GPS device is used during 9 days each and the travel diary is filled up during 8 days.
Changes in active commuting (classic or electric bike, public transport, walk, carpooling) from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  Active commuting will be measured by calculating the variables of interest from travel diary (kilometers traveled, modal share). The GPS device is used during 9 days each and the travel diary is filled up during 8 days.
Changes in active commuting (classic or electric bike, public transport, walk, carpooling) from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Active commuting will be measured using the GPS tracks and by calculating the variables of interest from travel diary (kilometers traveled, modal share). The GPS device is used during 9 days each and the travel diary is filled up during 8 days.
Changes in active commuting (classic or electric bike, public transport, walk, carpooling) from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  Active commuting will be measured by calculating the variables of interest from travel diary (kilometers traveled, modal share). The GPS device is used during 9 days each and the travel diary is filled up during 8 days.
Changes in minutes of moderate-to-vigorous physical activity (MVPA) from the baseline and and the beginning of the intervention (one month after the beginning of the intervention, Month 1) | Baseline and one month and a half after the baseline (Month 1)
  MVPA will be assessed by a tri-axial accelerometer (SenseDoc) with measurement frequency of 60 Hz during 9 days by the IPAQ (International Physical Activity Questionnaire) filled up once for the whole last week
Changes in minutes of moderate-to-vigorous physical activity (MVPA) from the baseline and the half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  MVPA will be assessed by a tri-axial accelerometer (SenseDoc) with measurement frequency of 60 Hz during 9 days by the IPAQ (International Physical Activity Questionnaire) filled up once for the whole last week
Changes in minutes of moderate-to-vigorous physical activity (MVPA) from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  MVPA will be assessed by a tri-axial accelerometer (SenseDoc) with measurement frequency of 60 Hz during 9 days by the IPAQ (International Physical Activity Questionnaire) filled up once for the whole last week
Changes in minutes of moderate-to-vigorous physical activity (MVPA) from the baseline and two months after the end of the intervention (Month 9) | Baseline, and nine months after the baseline (Month 9)
  MVPA will be assessed by the IPAQ (International Physical Activity Questionnaire) filled up once for the whole last week
Changes in minutes of moderate-to-vigorous physical activity (MVPA) from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  MVPA will be assessed by the IPAQ (International Physical Activity Questionnaire) filled up once for the whole last week
Changes in minutes of moderate-to-vigorous physical activity (MVPA) from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  MVPA will be assessed by a tri-axial accelerometer (SenseDoc) with measurement frequency of 60 Hz during 9 days by the IPAQ (International Physical Activity Questionnaire) filled up once for the whole last week
Changes in minutes of moderate-to-vigorous physical activity (MVPA) from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  MVPA will be assessed by the IPAQ (International Physical Activity Questionnaire) filled up once for the whole last week
Changes in exposure to air quality from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Exposure to air quality will be measured by the assessment of the concentration and composition of fine particles using a pollution captor (MicroPEMTM) during 8 days
Changes in exposure to air quality from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Exposure to air quality will be measured by the assessment of the concentration and composition of fine particles using a pollution captor (MicroPEMTM) during 8 days
Changes in self-reported quality of life from the baseline and the half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  Self-reported quality of life via questionnaire SF-12 (scale from 1 poor health to 5 good health)
Changes in self-reported quality of life from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  SSelf-reported quality of life via questionnaire SF-12 (scale from 1 poor health to 5 good health)
Changes in self-reported quality of life from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  Self-reported quality of life via questionnaire SF-12 (scale from 1 poor health to 5 good health)
Changes in self-reported quality of life from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  Self-reported quality of life via questionnaire SF-12 (scale from 1 poor health to 5 good health)
Changes in self-reported biometrics from the baseline and and the beginning of the intervention (one month after the beginning of the intervention, Month 1) | Baseline and one month and a half after the baseline (Month 1)
  Self-reported biometrics via biometric questionnaire
Changes in self-reported biometrics from the baseline and the half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  Self-reported biometrics via biometric questionnaire
Changes in self-reported biometrics from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Self-reported biometrics via biometric questionnaire
Changes in self-reported biometrics from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Self-reported biometrics via biometric questionnaire
Motivational stage from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Motivational stage via a Stage-of-change questionnaire (Biehl et al., 2018)
Motivational stage from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  Motivational stage via a Stage-of-change questionnaire (Biehl et al., 2018) (three questions that allow to classifie the people in precontemplation, contemplation, preparation, action, maintenance)
Motivational stage from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Motivational stage via a Stage-of-change questionnaire (Biehl et al., 2018) (three questions that allow to classifie the people in precontemplation, contemplation, preparation, action, maintenance)
Motivational stage from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  Motivational stage via a Stage-of-change questionnaire (Biehl et al., 2018) (three questions that allow to classifie the people in precontemplation, contemplation, preparation, action, maintenance)
Green self-identity from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Green self-identity via green self-identity (Lalot et al. 2019) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of green self-identity
Green self-identity from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  Green self-identity via green self-identity (Lalot et al. 2019) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of green self-identity
Green self-identity from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Green self-identity via green self-identity (Lalot et al. 2019) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of green self-identity
Green self-identity from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  Green self-identity via green self-identity (Lalot et al. 2019) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of green self-identity
Changes in habits of alternative modes to the car and car use from the baseline and and the beginning of the intervention (one month after the beginning of the intervention, Month 1) | Baseline and one month and a half after the baseline (Month 1)
  Habits of alternative modes to the car and car use via self-report habit index (Gardner et al., 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of habit
Changes in habits of alternative modes to the car and car use from the baseline and the half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  Habits of alternative modes to the car and car use via self-report habit index (Gardner et al., 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of habit
Changes in habits of alternative modes to the car and car use from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Habits of alternative modes to the car and car use via self-report habit index (Gardner et al., 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of habit
Changes in habits of alternative modes to the car and car use from the baseline and two months after the end of the intervention (Month 9) | Baseline, and nine months after the baseline (Month 9)
  Habits of alternative modes to the car and car use via self-report habit index (Gardner et al., 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of habit
Changes in habits of alternative modes to the car and car use from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  Habits of alternative modes to the car and car use via self-report habit index (Gardner et al., 2012)
Changes in habits of alternative modes to the car and car use from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Habits of alternative modes to the car and car use via self-report habit index (Gardner et al., 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of habit
Changes in habits of alternative modes to the car and car use from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  Habits of alternative modes to the car and car use via self-report habit index (Gardner et al., 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of habit
Changes in intention toward alternative modes to the car and car use from the baseline and and the beginning of the intervention (one month after the beginning of the intervention, Month 1) | Baseline and one month and a half after the baseline (Month 1)
  Intention toward alternative modes to the car and car use via intention questionnaire (Godin, 2012)
Changes in intention toward alternative modes to the car and car use from the baseline and the half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  Intention toward alternative modes to the car and car use via intention questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention
Changes in intention toward alternative modes to the car and car use from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Intention toward alternative modes to the car and car use via intention questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention
Changes in intention toward alternative modes to the car and car use from the baseline and two months after the end of the intervention (Month 9) | Baseline, and nine months after the baseline (Month 9)
  Intention toward alternative modes to the car and car use via intention questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention
Changes in intention toward alternative modes to the car and car use from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  Intention toward alternative modes to the car and car use via intention questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention
Changes in intention toward alternative modes to the car and car use from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Intention toward alternative modes to the car and car use via intention questionnaire (Godin, 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention
Changes in intention toward alternative modes to the car and car use from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  Intention toward alternative modes to the car and car use via intention questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention
Changes in self-efficacy for alternative modes and for the car from the baseline and and the beginning of the intervention (one month after the beginning of the intervention, Month 1) | Baseline and one month and a half after the baseline (Month 1)
  Self-efficacy for alternative modes and for the car via self-efficacy questionnaire (Schwarzer et al., 2015) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of self-efficacy
Changes in self-efficacy for alternative modes and for the car from the baseline and the half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  Self-efficacy for alternative modes and for the car via self-efficacy questionnaire (Schwarzer et al., 2015)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of self-efficacy
Changes in self-efficacy for alternative modes and for the car from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Self-efficacy for alternative modes and for the car via self-efficacy questionnaire (Schwarzer et al., 2015) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of self-efficacy
Changes in self-efficacy for alternative modes and for the car from the baseline and two months after the end of the intervention (Month 9) | Baseline, and nine months after the baseline (Month 9)
  Self-efficacy for alternative modes and for the car via self-efficacy questionnaire (Schwarzer et al., 2015) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of self-efficacy
Changes in self-efficacy for alternative modes and for the car from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  Self-efficacy for alternative modes and for the car via self-efficacy questionnaire (Schwarzer et al., 2015) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of self-efficacy
Changes in self-efficacy for alternative modes and for the car from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Self-efficacy for alternative modes and for the car via self-efficacy questionnaire (Schwarzer et al., 2015) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of self-efficacy
Changes in self-efficacy for alternative modes and for the car from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  Self-efficacy for alternative modes and for the car via self-efficacy questionnaire (Schwarzer et al., 2015) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of self-efficacy
Changes in intention implementation from the baseline and and the beginning of the intervention (one month after the beginning of the intervention, Month 1) | Baseline and one month and a half after the baseline (Month 1)
  Intention implementation via intention implementation questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention implementation
Changes in intention implementation from the baseline and the half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  Intention implementation via intention implementation questionnaire (Godin, 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention implementation
Changes in intention implementation from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Intention implementation via intention implementation questionnaire (Godin, 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention implementation
Changes in intention implementation from the baseline and two months after the end of the intervention (Month 9) | aseline, and nine months after the baseline (Month 9)
  Intention implementation via intention implementation questionnaire (Godin, 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention implementation
Changes in intention implementation from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  Intention implementation via intention implementation questionnaire (Godin, 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention implementation
Changes in intention implementation from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Intention implementation via intention implementation questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention implementation
Changes in intention implementation from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  Intention implementation via intention implementation questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of intention implementation
Changes in attitudes toward alternative modes to the car and toward car use from the baseline and and the beginning of the intervention (one month after the beginning of the intervention, Month 1) | Baseline and one month and a half after the baseline (Month 1)
  Attitudes toward alternative modes to the car and toward car use via attitudes questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of positive or negative attitudes
Changes in attitudes toward alternative modes to the car and toward car use from the baseline and the half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  Attitudes toward alternative modes to the car and toward car use via attitudes questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of positive or negative attitudes
Changes in attitudes toward alternative modes to the car and toward car use from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Attitudes toward alternative modes to the car and toward car use via attitudes questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of positive or negative attitudes
Changes in attitudes toward alternative modes to the car and toward car use from the baseline and two months after the end of the intervention (Month 9) | Baseline, and nine months after the baseline (Month 9)
  Attitudes toward alternative modes to the car and toward car use via attitudes questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of positive or negative attitudes
Changes in attitudes toward alternative modes to the car and toward car use from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  Attitudes toward alternative modes to the car and toward car use via attitudes questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of positive or negative attitudes
Changes in attitudes toward alternative modes to the car and toward car use from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Attitudes toward alternative modes to the car and toward car use via attitudes questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of positive or negative attitudes
Changes in attitudes toward alternative modes to the car and toward car use from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  Attitudes toward alternative modes to the car and toward car use via attitudes questionnaire (Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of positive or negative attitudes
Changes in perceived susceptibility and perceived severity of getting coronavirus disease from the baseline and and the beginning of the intervention (one month after the beginning of the intervention, Month 1) | Baseline and one month and a half after the baseline (Month 1)
  Perceived susceptibility and perceived severity of getting coronavirus disease via perceived risks questionnaire (Nexøe et al., 1999) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of perceived risks of getting COVID
Changes in perceived susceptibility and perceived severity of getting coronavirus disease from the baseline and the half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  Perceived susceptibility and perceived severity of getting coronavirus disease via perceived risks questionnaire (Nexøe et al., 1999)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of perceived risks of getting COVID
Changes in perceived susceptibility and perceived severity of getting coronavirus disease from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Perceived susceptibility and perceived severity of getting coronavirus disease via perceived risks questionnaire (Nexøe et al., 1999)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of perceived risks of getting COVID
Changes in perceived susceptibility and perceived severity of getting coronavirus disease from the baseline and two months after the end of the intervention (Month 9) | Baseline, and nine months after the baseline (Month 9)
  Perceived susceptibility and perceived severity of getting coronavirus disease via perceived risks questionnaire (Nexøe et al., 1999)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of perceived risks of getting COVID
Changes in perceived susceptibility and perceived severity of getting coronavirus disease from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  Perceived susceptibility and perceived severity of getting coronavirus disease via perceived risks questionnaire (Nexøe et al., 1999)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of perceived risks of getting COVID
Changes in perceived susceptibility and perceived severity of getting coronavirus disease from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Perceived susceptibility and perceived severity of getting coronavirus disease via perceived risks questionnaire (Nexøe et al., 1999)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of perceived risks of getting COVID
Changes in perceived susceptibility and perceived severity of getting coronavirus diseasefrom the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  Perceived susceptibility and perceived severity of getting coronavirus disease via perceived risks questionnaire (Nexøe et al., 1999)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of perceived risks of getting COVID
Changes in subjective norms toward alternative modes to the car and car use from the baseline and and the beginning of the intervention (one month after the beginning of the intervention, Month 1) | Baseline and one month and a half after the baseline (Month 1)
  Subjective norms toward alternative modes to the car and car use via subjective norms questionnaire(Godin, 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of subjective norms
Changes in subjective norms toward alternative modes to the car and car use from the baseline and the half of the intervention (Month 3) | Baseline, and three months after the baseline (Month 3)
  Subjective norms toward alternative modes to the car and car use via subjective norms questionnaire(Godin, 2012) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of subjective norms
Changes in subjective norms toward alternative modes to the car and car use from the baseline and the end of the intervention (Month 7) | Baseline, and seven month after the baseline (Month 7)
  Subjective norms toward alternative modes to the car and car use via subjective norms questionnaire(Godin, 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of subjective norms
Changes in subjective norms toward alternative modes to the car and car use from the baseline and two months after the end of the intervention (Month 9) | aseline, and nine months after the baseline (Month 9)
  Subjective norms toward alternative modes to the car and car use via subjective norms questionnaire(Godin, 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of subjective norms
Changes in subjective norms toward alternative modes to the car and car use from the baseline and six months after the end of the intervention (Month 12) | Baseline, and one year after the baseline (Month 12)
  Subjective norms toward alternative modes to the car and car use via subjective norms questionnaire(Godin, 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of subjective norms
Changes in subjective norms toward alternative modes to the car and car use from the baseline and one year after the end of the intervention (Month 18) | Baseline, and one year and a half after the baseline (Month 18)
  Subjective norms toward alternative modes to the car and car use via subjective norms questionnaire(Godin, 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of subjective norms
Changes in subjective norms toward alternative modes to the car and car use from the baseline and one year and a half after the end of the intervention (Month 24) | Baseline, and two years after the baseline (Month 24)
  Subjective norms toward alternative modes to the car and car use via subjective norms questionnaire(Godin, 2012)(scale from 1, Very much disagree and 7, strongly agree) to measure the strength of subjective norms
Changes in carbon footprint associated to transport | To be defined
  Carbon footprint associated to transport will be calculated considering the motorization (and type of car), kilometers traveled by car, and the use of alternative modes to the car

OTHER OUTCOMES:
Reach of the intervention | During the recruitment and enrollement, an average of 2 years
  Reach of the intervention via the calculation of the ratio of the participants contacted, eligible, and enrolled in the intervention
Quality of the implementation | During the implementation of the intervention, an average of 2 years
  Quality of the implementation via a checklist of al the tasks completed by the "mobility coach" (using a scale of yes or no)
Travel satisfaction | Baseline
  Travel satisfaction via satisfaction travel scale (Ettema et al. 2011) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of travel satisfaction
Autonomous and controlled motivation for alternative modes to the car | Month 0
  Autonomous and controlled motivation for alternative modes to the car via an adapted version of the motivation scale toward health-oriented physical activity (Boiché et al. 2019) (scale from 1, Very much disagree and 7, strongly agree) to measure the strength of autonomous motivation and controlled motivation
Accessibility and fluidity according to transport modes | Baseline
  Accessibility and fluidity according to transport modes via the calculation of spatial information associated with the place of residenc, place of work and the type of travel
Self-control ressources | Baseline
  Self-control ressources via the scale of availability of self-control resources (Ryan & Frederick, 1997) (scale from 1, Very much disagree and 7, strongly agree) to measure the amount of self-control ressources
Self-control ressources | One month and a half after the baseline (Month 1)
  Self-control ressources via the scale of availability of self-control resources (Ryan & Frederick, 1997) (scale from 1, Very much disagree and 7, strongly agree) to measure the amount of self-control ressources
Self-control ressources | Three months after the baseline (Month 3)
  Self-control ressources via the scale of availability of self-control resources (Ryan & Frederick, 1997) (scale from 1, Very much disagree and 7, strongly agree) to measure the amount of self-control ressources
Self-control ressources | Seven months after the baseline (Month 7)
  Self-control ressources via the scale of availability of self-control resources (Ryan & Frederick, 1997) (scale from 1, Very much disagree and 7, strongly agree) to measure the amount of self-control ressources
Self-control ressources | Nine months after the baseline (Month 9)
  Self-control ressources via the scale of availability of self-control resources (Ryan & Frederick, 1997) (scale from 1, Very much disagree and 7, strongly agree) to measure the amount of self-control ressources
Self-control ressources | One year after the baseline (Month 12)
  Self-control ressources via the scale of availability of self-control resources (Ryan & Frederick, 1997) (scale from 1, Very much disagree and 7, strongly agree) to measure the amount of self-control ressources
Self-control ressources | One year and a half after the baseline (Month 18)
  Self-control ressources via the scale of availability of self-control resources (Ryan & Frederick, 1997) (scale from 1, Very much disagree and 7, strongly agree) to measure the amount of self-control ressources
Self-control ressources | Two years after the baseline (Month 24)
  Self-control ressources via the scale of availability of self-control resources (Ryan & Frederick, 1997) (scale from 1, Very much disagree and 7, strongly agree) to measure the amount of self-control ressources

CONTACTS AND LOCATIONS:
Overall Officials: Aïna Chalabaev, Professor, Study Director — Laboratoire SENS, Univ. Grenoble-Alpes
Locations (1):
- Univ. Grenoble-Alpes, Saint-Martin-d'Hères, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Yes
Data dictionary, statistical analysis plan, informed consent form, analytic code will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study Protocole and informed consent form will be available in 2021, the clinical study report and the analytic code will be available after the end of the study (in 2025 or 2026)
Access Criteria: Study protocole preprint, informed consent form, clinical study report preprint and analytic code will be available on OSF platform for everybody
URL: http://osf.io/9anpg/

REFERENCES:
- [Derived] Teran-Escobar C, Duche S, Bouscasse H, Isoard-Gatheur S, Juen P, Lacoste L, Lyon-Caen S, Mathy S, Ployon E, Risch A, Sarrazin P, Slama R, Tabaka K, Treibich C, Chardonnel S, Chalabaev A. InterMob: a 24-month randomised controlled trial comparing the effectiveness of an intervention including behavioural change techniques and free transport versus an intervention including air pollution awareness-raising on car use reduction among regular car users living in Grenoble, France. BMC Public Health. 2022 Sep 16;22(1):1763. doi: 10.1186/s12889-022-14099-4. PMID 36114537